CLINICAL TRIAL: NCT03587454
Title: TELEGLAUCOMA: THE NJ HEALTH FOUNDATION STUDY a Prospective, Single Site, Masked Study Comparing the Diagnostic Accuracy and Management Recommendations of Teleglaucoma to Conventional Clinical Care in Patients With Glaucoma
Brief Title: Feasibility of Teleglaucoma Versus Conventional Clinical Evaluation for Diagnostic Accuracy and Management Recommendations in Patients With Glaucoma
Acronym: Teleglaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: New Jersey Health Foundation (Other)
Responsible Party: Principal Investigator, Albert S Khouri, MD, Associate Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Sequential | Purpose: Diagnostic
Other Study IDs: Pro20140001070
Record Dates: First submitted 2018-05-21; First posted 2018-07-16 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Teleglaucoma; Teleophthalmology; Glaucoma
Keywords: teleglaucoma; teleophthalmology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Prospective sequential enrolment in teleglaucoma then conventional glaucoma clinical care
Masking Description: Investigators in teleglaucoma and conventional glaucoma clinics are masked to one another
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-Glaucoma arm (Experimental): Subjects enrolled in tele-glaucoma arm for remote assessment
  Interventions: Diagnostic Test: Teleglaucoma

INTERVENTIONS:
Diagnostic Test: Teleglaucoma — Subjects are evaluated through a teleglaucoma protocol then by physical presence in a glaucoma clinic
  Other Names: teleophthalmology

SUMMARY:
Telemedicine allows screening of subjects with limited access to eye care. Failure of screenees to come for full examination was identified as a serious problem. Teleglaucoma should allow a single physician access to screenees in real time. The investigators aim to test the technical feasibility of developing a system for teleglaucoma that will allow a physician real time access to patient information and images and compare it to traditional physical presence evaluation in glaucoma clinics. This system can be applied during telemedicine for glaucoma and other vision threatening diseases.

DETAILED DESCRIPTION:
Research Plan including Methods

Investigators propose to develop a program for teleglaucoma and to validate it for patient care outcomes. The study will be conducted in two phases. The first phase will establish the technical foundation for the teleophthalmology system; the second phase will investigate the clinical impact of teleglaucoma.

Phase I: Investigators will develop and test technical aspects of a teleophthalmology system for glaucoma. Phase II will evaluate the impact of teleglaucoma on patient care outcomes.

Phase I. Development and Validation of a Teleophthalmology System in Glaucoma. By partnering with an ongoing telemedicine program at the Institute of Ophthalmology & Visual Science (IOVS), investigators will develop and test a system for telemedicine in glaucoma. In this phase, a wireless secure telemedicine system will be assembled that allows real-time access to participant subject screening data and images. The teleophthalmology system will be used and tested during telemedicine screening operations that are conducted by the investigators telemedicine team monthly in NJ. Telemedicine screenings occur all over the state of NJ at community centers, schools, places of worship, soup kitchens, other.

Telemedicine system component assembly: Integration to imaging equipment, setup, installation, and training of personnel will be performed.

In summary, this phase includes setup of imaging equipment (anterior segment and fundus camera) to the system, training of personnel, and post-installation quality checks by a communication technology expert. The server and specialized software will be customized for data entry, storage and display of selected patient health data in a secure configuration for internet access. Data obtained during routine IOVS telemedicine outreach program screening including demographic data, medical and ocular history, comprehensive ocular screening data (including imaging of the anterior and posterior ocular segments) will be configured for real time remote access by a physician. This phase also includes obtaining license to access a secure connection, and system configuration to allow data to be encrypted and securely transmitted using a Digital Imaging and Communications in Medicine (DICOM) format. Virtual storage of data will be configured, and monitors with visualization technology applications will be installed to communicate with the imaging devices used in telemedicine.

During this phase quality measures will be tracked, recorded and analyzed. Those system quality checks will include 1. quality of acquired and transmitted ocular images (exposure, color, focus, etc.) 2. data security (Digital Imaging and Communications in Medicine encryption) 3. speed of data transmission (real-time network streamlining, interruptions and delays) obtained during each testing session.

Phase II. Patient Outcomes: Teleglaucoma vs Conventional Care

A population of patients seeking glaucoma care at IOVS glaucoma clinics will be included in this phase of the study. Subjects will be enrolled over a 6 month period. Subjects referred to or who are established patients at IOVS' glaucoma clinics will be enrolled on the same day in the teleglaucoma screening program and glaucoma clinic (physical presence). Two glaucoma fellowship-trained physician investigators will perform diagnostic and therapeutic recommendations during teleglaucoma and in glaucoma clinics. Participant patients will go through the consent process. All questions about the study will be explained by investigators. Upon consent process completion the participant will first undergo testing through the telemedicine protocol (see below). Data and images will then be transmitted. The investigator physician evaluating teleglaucoma data will assess the patient data and a diagnosis, management and follow-up recommendation will be made. The participant subject will then proceed to glaucoma clinic, where the participant will be examined by the investigator physician in the glaucoma clinic according to standard of care practices. The investigator physician physically present in the glaucoma clinics and the investigator physician in the teleglaucoma reading room will be masked to each other's recommendations regarding diagnostic tests and therapeutic recommendations.

Data regarding the accuracy of diagnostic tests (e.g., visual acuity, tonometry, optic nerve assessment, and other routine glaucoma tests) from teleglaucoma and from physical presence will be compared. The accuracy of glaucoma diagnosis (no glaucoma, glaucoma suspect, confirmed Glaucoma) and management recommendations will also be compared. Parameters to be studied will include comparisons of LogMAR visual acuity, tonometry, ocular examination and particularly optic nerve evaluation (estimation of vertical and horizontal cup-to-disc ratio, presence of signs of glaucomatous neuropathy: disc hemorrhage, notching, localized pallor, and asymmetry in cup-to-disc ratio of the two eyes >0.2 disc diameters, among others). Limitations to an adequate ocular examination or imaging during teleglaucoma and physical presence will be tracked. Inter-observer agreement between the two arms (teleglaucoma and physical presence) will be determined.

The accuracy of glaucoma diagnosis, i.e., confirmed glaucoma, glaucoma suspect, no glaucoma, as well as management recommendations, i.e., monitoring care, therapeutic interventions, obtained via teleglaucoma and physical presence will be compared. Statistical analyses will be performed on collected data. All data will be collected by subject codes. No protected health information will be gathered. Statistical analysis will be performed using statistical software through consultation with a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with glaucoma or who are glaucoma suspects

Exclusion Criteria:

* Physical limitations precluding image acquisition like the inability to position for imaging or the inability to acquire images/testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of diagnosis and management in Teleglaucoma and conventional care | 24 months
  Qualitative categorical outcome:
  Glaucoma Diagnosis, Management and follow up are clinical determinations by the investigator that are based on the overall clinical evaluation of the subject
  Diagnosis: A. no glaucoma B. confirmed glaucoma
  Management: A. maintain current therapy, B. advance therapy (additional glaucoma medication or surgical glaucoma intervention), C. no therapy needed
  Follow up: A. urgent (less than 4 weeks from time of evaluation) B. routine (more than 4 weeks from time of evaluation)

SECONDARY OUTCOMES:
Assessment of diagnostic tools during teleglaucoma: Visual acuity | 12 months
  Quantitative outcome:
  Visual Acuity will be measured on the Snellen chart and then converted to a Log MAR scale (Logarithm of the Minimal Angle of Resolution scale= Log MAR scale). Log MAR scale:
  0.0 to 2.0 units (in increments of 0.2) with 0.0 units representing 20/20 visual acuity (normal vision) and higher numbers representing worse visual acuity (2.0 units representing poor vision of 20/2000)
Assessment of diagnostic tools during teleglaucoma: Tonometry | 12 months
  Quantitative outcome:
  Tonometry will be measured using a Goldmann applanation tonometer and a puff tonometer. All measurements will be in mm Hg, range 0.0-60.0 mm Hg (in increments of 1 mm Hg). Normal range is 6-21 mm Hg. Measurements below 6 and above 21 mm Hg are considered outside the normal range.
Assessment of diagnostic tools during tele glaucoma: Optic nerve | 12 months
  Quantitative outcome:
  Vertical and Horizontal cup-to-disc rations 0.0-1.0 (in increments of 0.1) will be measured. Ratio>0.6 are considered higher risk for glaucoma.
  All measurements will be made by investigators on a high resolution monitor in a dark room. Investigators will be masked to one another assessments in instances were multiple readings are obtained. Images will be presented in a random order when multiple measures are obtained. Other Anterior and posterior segment pathology will be qualitatively noted (cataract, narrow angle, cornea pathology, diabetic retinopathy, age related macular degeneration, other).
Assessment of diagnostic tools during tele glaucoma: Optical Coherence Tomography | 12 months
  Quantitative outcome:
  Optical Coherence Tomography (OCT) will be used to obtain images of the anterior and posterior ocular segments.
  Quantitative measures in micron: 0-900 micron (+/- 5 micron) will be recorded for the cornea, optic nerve and retina. The range of normal is based on reference data that is age and racially determined.

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Khouri, MD, Principal Investigator — Rutgers University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandrasekaran S, Kass W, Thangamathesvaran L, Mendez N, Khouri P, Szirth BC, Khouri AS. Tele-glaucoma versus clinical evaluation: The New Jersey Health Foundation Prospective Clinical Study. J Telemed Telecare. 2020 Oct;26(9):536-544. doi: 10.1177/1357633X19845273. Epub 2019 May 28. PMID 31138016